CLINICAL TRIAL: NCT06681181
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Target Engagement of GSK4528287 in Healthy Participants
Brief Title: A First-time in Human (FTIH) Study to Evaluate Safety, Tolerability, Pharmacokinetics and Target Engagement of GSK4528287 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221603
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Colitis, Ulcerative
Keywords: Inflammatory bowel disease; Crohns disease; Ulcerative colitis; GSK4528287; First time in human (FTIH); Healthy participants; GlaxoSmithKline (GSK)
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is single centre, double-blind study.
Who Masked: Participant, Investigator
Masking Description: The investigators will be blinded not knowing which study intervention each participant will be assigned to and this will be maintained throughout the course of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1: Dose 1 (Experimental): Participants will be administered Dose 1 of GSK4528287.
  Interventions: Drug: GSK4528287
- Cohort 2: Dose 2 (Experimental): Participants will be administered Dose 2 of GSK4528287.
  Interventions: Drug: GSK4528287
- Cohort 3: Dose 3 (Experimental): Participants will be administered Dose 3 of GSK4528287.
  Interventions: Drug: GSK4528287
- Cohort 4: Dose 4 (Experimental): Participants will be administered Dose 4 of GSK4528287.
  Interventions: Drug: GSK4528287
- Cohort 5: Dose 5 (Experimental): Participants will be administered Dose 5 of GSK4528287.
  Interventions: Drug: GSK4528287
- Cohort 6: Dose 6 (Experimental): Participants will be administered Dose 6 of GSK4528287.
  Interventions: Drug: GSK4528287
- Placebo (Placebo Comparator): Participants will receive Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK4528287 — GSK4528287 will be administered.
  Arms: Cohort 1: Dose 1; Cohort 2: Dose 2; Cohort 3: Dose 3; Cohort 4: Dose 4; Cohort 5: Dose 5; Cohort 6: Dose 6
Drug: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
"GSK4528287 is a drug being developed to treat like inflammatory bowel diseases like Crohns disease and ulcerative colitis. This study is the first time that GSK4528287 will be given to humans. The study will test single doses of GSK4528287 to check for side effects, measure blood levels, and understand how it works in the body. The study will start with a small dose, and the dose will be increased for each new group of participants."

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* White blood cell greater than or equal to (>=) lower limit of normal (LLN), including both lymphocyte counts >= LLN and neutrophil counts >= LLN, at both screening and pre-dose (Day-1) Note: in cases where the test is abnormal, the participant may have the test repeated once and if their second test is normal, they will be eligible. In the event a second test is also abnormal, the participant is not eligible
* Electrocardiogram (ECG) with no clinically significant abnormality at the discretion of the investigator/designee
* Participants with a confirmed positive vaccination status for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines as per local/site guidance
* SARS-CoV-2 screening test negative as per local guidance
* If dosing is during influenza season (October to April per local guidelines), participants who have not had a seasonal influenza vaccine must receive a medicines and healthcare products regualtory agency (MHRA)-approved influenza vaccine at least 30 days before dosing
* Body weight >= 50 kilograms (kg) and body mass index (BMI) within the range 18-32 kilograms per square meters (kg/m^2) (inclusive)
* Male and/or female of non-childbearing potential
* Male participants are eligible to participate if they agree to the following during the study intervention period and for 48 weeks after the single dose of study intervention: refrain from donating sperm; be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant
* A female participant is eligible to participate if she is a woman of non-childbearing potential (WONCBP)
* Capable of giving signed informed consent

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data
* Abnormal blood pressure as determined by the investigator
* Symptomatic herpes zoster within 3 months prior to screening
* Prior medical history of anaphylaxis or severe adverse reactions to vaccines
* Significant allergies to humanized monoclonal antibodies
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear Immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Immunodeficiency or autoimmunity assessed by medical history.
* A history of recurrent infections
* Treatment of any significant infection within 3 months prior to the first dose of study drug, including both serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, shingles)
* Any history of chronic infection including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Any acute infection (including upper respriatory tract infection [URTI] and urinary tract infection [UTI]) which has not fully resolved within four weeks of dosing
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) medical monitor, poses a safety risk with regards to participation in the trial
* History of malignancy, including malignant or non-malignant skin cancer
* Prior moderate/severe SARS-CoV-2 infection requiring oxygen supplementation or admission to hospital
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Antibiotics or antiviral therapy within 30 days of dosing
* Receipt of live vaccination within 1 month prior to screening or plan to receive live vaccination during the study
* Past or intended use of over the counter or prescription medication including herbal medications within 7 days prior to dosing
* The participant has participated in a clinical trial and has received an investigational product (IP) within the following time-period prior to the first dosing day of the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than 4 new chemical entities within 12 months prior to dosing
* Current enrolment or past participation in this clinical study.
* Participation in a clinical study that would result in donation of blood or blood products in excess of 500 millilitres (mL) within a 56 day period
* A positive diagnostic Mycobacterium tuberculosis bacteria (MTB) test at screening (defined as positive QuantiFERON Gold test)
* Positive test for HIV antibody at screening
* Positive drug/alcohol test, including tetrahydrocannabinol, at screening or Day 1
* Positive smoke breath analyzer levels indicative of smoking history at screening and in house admission to the clinical research unit or regular use of tobacco- or nicotine-containing products (e.g., nicotine patches, vaporizing devices) within 6 months prior to screening
* A positive confirmation of SARS CoV 2 infection or signs and symptoms suggestive of SARS CoV 2 at screening or pre dose
* The participant is at high risk of MTB infection in the opinion of the Investigator. Risk factors include residing in a high prevalence area or having close contact with a person with confirmed MTB infection
* The participant has a phobia to needles
* Regular alcohol consumption within 6 months prior to study, defined as: An average weekly intake of greater than (>)14 units of alcohol. One unit is equivalent to 8 grams (g) of alcohol: a half pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits
* Regular use of known drugs of abuse, including tetrahydrocannabinol
* Alanine aminotransferase (ALT or AST) >1.0*upper limit of normal (ULN)
* Total bilirubin >1.0*ULN; Participants with Gilbert's syndrome can be included with total bilirubin >1.5*ULN as long as direct bilirubin is less than or equal to (<=) 1.5*ULN
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at screening or Day -1 or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* QTcF (QT interval corrected for heart rate according to Fredericia's formula) >450 milliseconds (msec).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2027-03-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Day 351 (End of follow up period)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of Participants with Serious Adverse Events (SAE) | Up to Day 351 (End of follow up period)
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: Results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant.
Number of Participants with Clinically Significant Changes in Laboratory Values | Up to Day 351 (End of follow up period)
  Number of participants with clinically significant changes in laboratory values (hematology, chemistry, urinalysis, and virology) will be assessed.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 351 (End of follow up period)
  Number of participants with clinically significant changes in vital signs will be assessed.
Number of Participants with Clinically Significant Changes in Telemetry | On Day 1
  Number of participants with clinically significant changes in telemetry will be assessed.
Number of Participants with Clinically Significant Changes in 12 lead Electrocardiogram (ECG) | Up to Day 351 (End of follow up period)
  Number of participants with clinically significant changes in 12 lead ECG will be assessed.

SECONDARY OUTCOMES:
Area under concentration-time curve (AUC) of GSK4528287 | Up to Day 337
  Blood sample will be collected to evaluate plasma concentration of AUC of GSK4528287.
Maximum concentration (Cmax) of GSK4528287 | Up to Day 337
  Blood sample will be collected to evaluate plasma concentration of Cmax of GSK4528287.
Time to maximum concentration (Tmax) of GSK4528287 | Up to Day 337
  Blood sample will be collected to evaluate plasma concentration of Tmax of GSK4528287.
Apparent terminal phase half life (T-half) of GSK4528287 | Up to Day 337
  Blood sample will be collected to evaluate plasma concentration of T-half of GSK4528287.
Clearance (CL) of GSK4528287 | Up to Day 337
  Blood sample will be collected to evaluate plasma concentration of CL of GSK4528287.
Bioavailability of GSK4528287 | Up to Day 337
  Blood sample will be collected to evaluate plasma concentration of SC bioavailability of GSK4528287.
Number of Participants with Confirmed Positive and Negative anti-GSK4528287 Antibodies | Up to Day 211
  Number of participants with confirmed positive and negative anti-GSK4528287 Antibodies will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/